CLINICAL TRIAL: NCT04470713
Title: Natural History Study for Pediatric Patients With Early Onset of Either GM1 Gangliosidosis, GM2 Gangliosidoses, or Gaucher Disease Type 2
Acronym: RETRIEVE
Status: Completed | Type: Observational
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-085A301; 2019-01125 (Other: BASEC)
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: GM1 Gangliosidosis; GM2 Gangliosidosis; Gaucher Disease, Type 2; Tay-Sachs Disease; AB Variant Gangliosidosis GM2; Sandhoff Disease
MeSH Terms: conditions — Gangliosidosis, GM1; Gangliosidoses, GM2; Gaucher Disease; Tay-Sachs Disease; Tay-Sachs Disease, AB Variant; Sandhoff Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A - Retrospective data collection: Participants with a confirmed diagnosis, either deceased patients or patients whose survival status is not known at enrollment.
- Group B - Prospective data collection: Participants who are alive at enrollment. Data collection is retrospective for the time between birth and enrollment visit, and data collection is prospective from the enrollment visit onwards. Visits are performed as per local standard of care.

SUMMARY:
This study is being conducted to better understand the natural course of GM1 gangliosidosis, GM2 gangliosidoses and Gaucher disease Type 2 (GD2). Information is planned to be gathered on at least 180 patients with GM1 gangliosidosis, GM2 gangliosidoses, and Gaucher Disease type 2. Retrospective data collection is planned for at least 150 deceased patients (Group A). Group B is for patients alive at the time of enrollment. In Group B it is planned to prospectively collect more comprehensive data from at least 30 patients. The purpose of this study is to collect relevant information for a adequate design of a potential subsequent research program in these diseases.

In this study no therapy is being offered.

ELIGIBILITY:
Inclusion Criteria:

* Patient with either GM1 gangliosidosis, GM2 gangliosidoses (Tay-Sachs, Sandhoff, or AB Variant), or Gaucher Disease Type 2.
* Diagnosis confirmed by either biochemical (enzyme activity) or genetic testing, or both.
* Date of birth on or after 1 January 2000.
* Onset of first neurological symptom within 24 months of age.
* Informed consent of parent or legal guardian as required by local law.

Min Age: 0 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted in hospitals/clinical centers managing pediatric patients with GM1 gangliosidosis, GM2 gangliosidoses, and/or Gaucher Disease type 2 across several countries in North America, South America, and Europe. In order to minimize the patient/data selection bias, the centers are asked to include all eligible patients from their center.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Survival of pediatric patients with early onset of GM1 gangliosidosis, GM2 gangliosidoses, and Gaucher Disease type 2 | 2.5 years

OTHER OUTCOMES:
Epidemiological data available from medical records | 2.5 years
  Patients' medical record data such as date of diagnosis, the date of appearance of first neurological symptom, dates of gain or loss of specific abilities (e.g. ability to sit) will be collected, if available.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (17):
- United States (3):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Lysosomal and Rare Disorders Research and Treatment Center, Fairfax, Virginia
- UCL Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Hospital de Clínicas de Porto Alegre - HCPA, Porto Alegre, Brazil
- AP-HP - Hôpitaux Universitaires Est Parisien, Paris, France
- SphinCS GmbH, Höchheim, Germany
- Italy (2):
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan
- Portugal (2):
  - Centro Hospitalar Universitario Lisboa Norte, EPE, Lisbon
  - Centro Universitario Hospitalar de São João, EPE, Porto
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Quirónsalud, Zaragoza
- Switzerland (2):
  - Universitätsspital Bern Inselspital, Bern
  - Universitäts-Kinderspital Zürich, Zurich
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Great Ormond Street Hospital for Children NHS Found. Trust, London

IPD SHARING:
Plan to Share IPD: No